CLINICAL TRIAL: NCT02784821
Title: Antibiotic Effects on the Developing Microbiome, Metabolome and Morbidities in Preterm Neonates
Brief Title: Antibiotic "Dysbiosis" in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Society for Pediatric Dermatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201501045-N; R21HD088005 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-27 (Estimated); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Enterocolitis, Necrotizing; Bacteremia; Bronchopulmonary Dysplasia; Intraventricular Hemorrhage; Periventricular Leukomalacia; Chronic Lung Disease; Ileal Perforation
MeSH Terms: conditions — Enterocolitis, Necrotizing; Bacteremia; Bronchopulmonary Dysplasia; Leukomalacia, Periventricular | interventions — Anti-Bacterial Agents; Ampicillin; Gentamicins; Cefotaxime; Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A - Antibiotics Indicated (Other): These neonates have a clinical indication to receive antibiotics such as symptoms out of expected for gestation OR delivered to moms with high perinatal infectious risks.
  The standard of care antibiotics include Ampicillin and Gentamicin or Cefotaxime.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Interventions: Drug: Antibiotic; Other: Gastric fluid; Other: Breast milk; Other: Stool samples
- Group B - antibiotics not indicated (Other): These neonates are asymptomatic AND are delivered to moms with low perinatal infectious risk factors.
  Antibiotics is not indicated for this group as standard of care.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Interventions: Other: Gastric fluid; Other: Breast milk; Other: Stool samples
- Group CI/randomized to antibiotics (Other): This group will be randomized to receive standard of care antibiotics which include Ampicillin and Gentamicin or Cefotaxime.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Interventions: Other: Gastric fluid; Other: Breast milk; Other: Stool samples; Drug: Antibiotics
- Group CII/randomized to no antibiotics (Other): This group will be randomized not to receive standard of care antibiotics.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Interventions: Other: Gastric fluid; Other: Breast milk; Other: Stool samples

INTERVENTIONS:
Drug: Antibiotic — Babies that are assigned to antibiotics receive therapy based on the clinical team's discretion.
  Other Names: Ampicillin or Gentamicin or Cefotaxime
  Arms: Group A - Antibiotics Indicated
Other: Gastric fluid — Microbiome evaluated using gastric aspirate.
  Other Names: Gastric aspirate
Other: Breast milk — Microbiome will be evaluated using mother's breast milk.
Other: Stool samples — Microbiome will be evaluated using infant's stool.
Drug: Antibiotics — Babies that are randomized to antibiotics receive therapy based on the clinical team's discretion.
  Other Names: Ampicillin or Gentamicin or Cefotaxime
  Arms: Group CI/randomized to antibiotics

SUMMARY:
Prolonged antibiotic use in preterm neonates has significant consequences on the developing intestinal microbiome, metabolome and host response, predisposing the neonate to various major morbidities, including necrotizing enterocolitis (NEC), late-onset sepsis, bronchopulmonary dysplasia (BPD), and mortality.

The hypothesis is that early and prolonged antibiotic use in preterm neonates has significant consequences on the developing intestinal microbiome, metabolome and host response, predisposing the neonate to various major morbidities. It is possible that the effect of this widespread antibiotic use outweighs the potential benefits. This study will randomize preterm infants born at less than 33 weeks gestation to either pre-emptive antibiotics or no-pre-emptive antibiotics.

The purpose of this research is to evaluate the risks and benefits of current practice to determine optimal levels of antibiotic use that protects the babies from infection with minimal effect on the microbiome and subsequent adverse outcomes related to overuse of antibiotics.

DETAILED DESCRIPTION:
A majority of preterm very low birthweight (VLBW) infants are exposed to antibiotics. Surveys from large databases in the US show that the rate of culture proven bacteremia in these infants at birth is only between 1-2 percent.

Antibiotic use, especially when repeated, induces a perturbation ("dysbiosis") in gut microbiota that may not recover to the basal state. Antibiotic use increases the risk of subsequent disease and adverse outcomes. The dependence of the developing immune system on the intestinal microbiota is supported by emerging evidence from studies in animals demonstrating decreased resistance to subsequent disease with early exposure to antibiotics.

A retrospective review of 50,0261 neonates across 127 neonatal intensive care units (NICUs) from California showed a forty-fold variation in NICU antibiotic prescribing practice with similar burdens of proven infection and mortality. A large number of preterm infants are thus subjected to a potentially harmful course of antibiotics that provides no clear benefit. There remains a major gap in our understanding of antibiotic-related intestinal microbial dysbiosis and how this may result in disease.

There will be two aims. In the first aim, a prospective, randomized pilot study, will test the effects of pre-emptive postnatal antibiotics on the microbiome, metabolome and inflammatory responses in the neonate during the NICU course. The second aim will assess the effects of pre-emptive postnatal antibiotics on adverse outcomes in the neonate while in the NICU. The hypothesis is that higher antibiotic use will not be associated with decreased early onset sepsis and in fact, will be associated with increased adverse outcomes including retinopathy of prematurity, necrotizing enterocolitis, spontaneous ileal perforation, late onset sepsis, chronic lung disease, bronchopulmonary dysplasia, intraventricular hemorrhage, periventricular leukomalacia, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All infants less than 33 weeks gestation.

Exclusion Criteria:

* Infants who are non-viable at birth.

Ages: 23 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Neu, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ojeda A, Akinsuyi O, McKinley KL, Xhumari J, Triplett EW, Neu J, Roesch LFW. Increased antibiotic resistance in preterm neonates under early antibiotic use. mSphere. 2024 Oct 29;9(10):e0028624. doi: 10.1128/msphere.00286-24. Epub 2024 Oct 7. PMID 39373498
- [Derived] Singh NK, Will L, Al-Mulaabed S, Ruoss L, Li N, de La Cruz D, Gurka M, Neu J. Antibiotics Use and Its Effects on the Establishment of Feeding Tolerance in Preterm Neonates. Am J Perinatol. 2024 May;41(S 01):e2248-e2253. doi: 10.1055/a-2108-1960. Epub 2023 Jun 12. PMID 37308133
- [Derived] Russell JT, Lauren Ruoss J, de la Cruz D, Li N, Bazacliu C, Patton L, McKinley KL, Garrett TJ, Polin RA, Triplett EW, Neu J. Antibiotics and the developing intestinal microbiome, metabolome and inflammatory environment in a randomized trial of preterm infants. Sci Rep. 2021 Jan 21;11(1):1943. doi: 10.1038/s41598-021-80982-6. PMID 33479274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study protocol was approved by the University of Florida IRB in September 2016. Enrollment occurred between January 2017 and January 2019. The study was paused for a full IRB review secondary to adverse outcomes and resumed when the incident of adverse outcomes was similar to the national standard.
  Actual enrollment was 98 infants.
Pre-assignment Details: 98 infants were enrolled in the study and were included in the arms of the study to receive intervention.
Groups:
- Group B: Antibiotics Not Indicated: Infant not receiving antibiotics secondary to asymptomatic and delivered to mom's without high perinatal infectious risk factors.
- Group A: Antibiotics Indicated: Infants delivered to high infectious risk mothers or infants with symptoms out of proportion to what is expected for gestational age.
- Group CI/Randomized to Antibiotics: Infants in Group CI/antibiotics were randomized to antibiotics.
  Infants were eligible for randomization if they were delivered to moms with low perinatal infectious risk factor AND they had symptoms as expected for gestation.
- Group CII/Randomized to no Antibiotics: Group CII/no antibiotics.
  Infant in group CII were randomized to no antibiotics.
  Infants were eligible for randomization if they were delivered to moms with low perinatal infectious risk factor AND they had symptoms as expected for gestation.
Period: Overall Study
Arm/Group | Group B: Antibiotics Not Indicated | Group A: Antibiotics Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Started | 11 | 32 | 28 | 27
Completed | 11 | 27 | 24 | 22
Not Completed | 0 | 5 | 4 | 5
Not completed — Death | 0 | 5 | 4 | 5

BASELINE CHARACTERISTICS:
Population: x2 test or ANOVA
Groups:
- Group A/Antibiotics Indicated: These neonates have a clinical indication to receive antibiotics, such as maternal chorioamnionitis with fetal tachycardia. The standard of care antibiotics include Ampicillin and Gentamicin or Cefotaxime and as part of standard of care blood tests such as complete blood cell counts, blood cultures, and C-reactive proteins will be performed.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Antibiotic: Babies that are assigned to antibiotics receive therapy based on the clinical team's discretion.
  Gastric fluid: Microbiome and inflammatory mediators will be evaluated using gastric aspirate.
  Breast milk: Microbiome, and inflammatory mediators will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
- Group B/Antibiotics Not Indicated: These neonates show no signs of respiratory distress(RDS) or have no indications of maternal chorioamnionitis. Antibiotics is not indicated for this group as standard of care.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Gastric fluid: Microbiome will be evaluated using gastric aspirate.
  Breast milk: Microbiome, metabolome, and inflammatory mediators will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
- Group CI/Randomized to Antibiotics: This group will be randomized to receive standard of care antibiotics which include Ampicillin and Gentamicin or Cefotaxime.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Gastric fluid: Microbiome will be evaluated using gastric aspirate.
  Breast milk: Microbiome will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
  Antibiotics - Babies that are randomized to antibiotics receive therapy based on the clinical team's discretion.
- Group CII/Randomized to no Antibiotics: This group will be randomized not to receive standard of care antibiotics. Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Gastric fluid: Microbiome will be evaluated using gastric aspirate.
  Breast milk: Microbiome will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
- Total: Total of all reporting groups
Arm/Group | Group A/Antibiotics Indicated | Group B/Antibiotics Not Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics | Total
Number analyzed (Participants) | 32 | 11 | 28 | 27 | 98
Age, Continuous [Mean (Standard Deviation); unit: gestation age in weeks]
  Gestational age | 28.2 (2.9) | 32.1 (1) | 29.2 (2.5) | 28.8 (2.8) | 29.1 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 15 | 10 | 48
  Male | 16 | 4 | 13 | 17 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 11 | 28 | 27 | 98
cesarean delivery [Count of Participants; unit: Participants] | 19 | 3 | 17 | 19 | 58
singleton [Count of Participants; unit: Participants] | 24 | 10 | 20 | 21 | 75
birth weight [Mean (Standard Deviation); unit: grams] | 1138 (446) | 1900 (417) | 1234 (424) | 1098 (384) | 1240 (479)

OUTCOME MEASURES:

1. Primary Outcome: Number of Events of Composite Morbidities and Mortality, Including Necrotizing Enterocolitis (NEC), Late Onset Sepsis (LOS), Bronchopulmonary Dysplasia (BPD) and Death
Description: Enrolled subjects' medical record will be reviewed to determine the number of patients with the composite outcome and the association between antibiotic administration and the components of the composite outcome
Time Frame: Until discharge from the NICU, up to 1 year
Measure: Number; unit: adverse events composite outcome
Groups:
- Group A/Antibiotics Indicated: These neonates have a clinical indication to receive antibiotics, such as maternal chorioamnionitis with fetal tachycardia. The standard of care antibiotics include Ampicillin and Gentamicin or Cefotaxime.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Antibiotic: Babies that are assigned to antibiotics receive therapy based on the clinical team's discretion.
  Gastric fluid: Microbiome will be evaluated using gastric aspirate.
  Breast milk: Microbiome will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
- Group B/Antibiotics Not Indicated: These neonates show no signs of respiratory distress(RDS) or have no indications of maternal chorioamnionitis. Antibiotics is not indicated for this group as standard of care.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Gastric fluid: Microbiome will be evaluated using gastric aspirate.
  Breast milk: Microbiome will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
- Group CI/ Randomized to Antibiotics: This group will be randomized to receive standard of care antibiotics which include Ampicillin and Gentamicin or Cefotaxime.
  Study interventions will include the collection of samples for the following: breast milk, gastric fluid and stool samples for analysis of the microbiome.
  Gastric fluid: Microbiome will be evaluated using gastric aspirate.
  Breast milk: Microbiome will be evaluated using mother's breast milk.
  Stool samples: Microbiome will be evaluated using infant's stool.
  Antibiotics: Babies that are randomized to antibiotics receive therapy based on the clinical team's discretion.
Arm/Group | Group A/Antibiotics Indicated | Group B/Antibiotics Not Indicated | Group CI/ Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Number analyzed (Participants) | 32 | 11 | 28 | 27
adverse events composite outcome | 19 | 1 | 9 | 14

2. Secondary Outcome: Number of Participants With Late Onset Sepsis
Description: Enrolled subjects' medical record will be reviewed to determine the number of patients who developed bacteremia after the first week of life (late onset sepsis) and the association between antibiotic administration and the development of late onset sepsis.
Time Frame: Until discharge from the NICU, up to 1 year
Population: x2 test
Measure: Number; unit: participants
Arm/Group | Group A: Antibiotics Indicated | Group B: Antibiotics Not Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Number analyzed (Participants) | 32 | 11 | 28 | 27
participants | 6 | 0 | 5 | 4

3. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD)
Description: Enrolled subjects' medical record will be reviewed to determine the number of patients who developed BPD and the association between antibiotic administration and diagnosis of BPD.
Time Frame: Until discharge from the NICU, up to 1 year
Population: x2 test
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Antibiotics Indicated | Group B: Antibiotics Not Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Number analyzed (Participants) | 32 | 11 | 28 | 27
Participants | 12 | 1 | 3 | 8

4. Secondary Outcome: Number of Participants With Necrotizing Enterocolitis (NEC)
Description: Enrolled subjects' medical record will be reviewed to determine the number of patients who developed NEC and the association between antibiotic administration and necrotizing enterocolitis
Time Frame: Until discharge from the NICU, up to 1 year
Population: x2 test
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Antibiotics Indicated | Group B: Antibiotics Not Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Number analyzed (Participants) | 32 | 11 | 28 | 27
Participants | 1 | 0 | 2 | 1

5. Secondary Outcome: Number of Deaths
Description: Enrolled subjects' medical record will be reviewed to determine the number of death prior to discharge from neonatal intensive care unit
Time Frame: until discharge from the NICU, up to one year.
Population: x2 test
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Antibiotics Indicated | Group B: Antibiotics Not Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Number analyzed (Participants) | 32 | 11 | 28 | 27
Participants | 5 | 0 | 4 | 5

6. Secondary Outcome: Length of Stay.
Description: length of stay in NICU in days.
Time Frame: Average days +/- standard deviation of hospitalization, up to 15 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group B: Antibiotics Not Indicated | Group A: Antibiotics Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
Number analyzed (Participants) | 11 | 32 | 28 | 27
days | 26.5 (19.7) | 64.5 (40.5) | 53.9 (30) | 61.6 (40.1)

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Group A: Antibiotics Indicated | Group B: Antibiotics Not Indicated | Group CI/Randomized to Antibiotics | Group CII/Randomized to no Antibiotics
All-Cause Mortality (participants affected / at risk) | 5/32 | 0/11 | 4/28 | 5/27
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/11 | 0/28 | 1/27
Other Adverse Events (participants affected / at risk) | 6/32 | 0/11 | 5/28 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Antibiotics Indicated (N=32) | Group B: Antibiotics Not Indicated (N=11) | Group CI/Randomized to Antibiotics (N=28) | Group CII/Randomized to no Antibiotics (N=27)
early onset sepsis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Antibiotics Indicated (N=32) | Group B: Antibiotics Not Indicated (N=11) | Group CI/Randomized to Antibiotics (N=28) | Group CII/Randomized to no Antibiotics (N=27)
late onset sepsis (Infections and infestations) | 6 (6) | 0 (0) | 5 (5) | 4 (4)

LIMITATIONS AND CAVEATS:
Limitations of our study are a small n, infants enrolled at the peri-viable and high risk gestation (high risk for mortality and serious adverse events), and high number of infants changed from group CII/no antibiotics to receive antibiotics in the first 48hours of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02784821/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02784821/ICF_002.pdf